CLINICAL TRIAL: NCT04111406
Title: Comparison of the Incidence of Inadequate Epidural Analgesia Between Protocol Based and Current Practice
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: covid19 situation
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: Si 342/2018
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Epidural Analgesia; Postoperative Pain
Keywords: Epidural Analgesia; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Historical control study (Before and after study) Data in current practice was derived from acute pain record before Jan 2019
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current practice (Other): Epidural insertion and epidural drug administration depend on anesthetist in charge
  Interventions: Drug: Current practice
- Protocol based (Experimental): Epidural insertion and epidural drug administration depend on anesthetist in research team using protocol based
  Interventions: Drug: Protocol based

INTERVENTIONS:
Drug: Current practice — Epidural insertion and epidural drug administration depend on anesthetist in charge
  Arms: Current practice
Drug: Protocol based — Epidural insertion and epidural drug administration depend on anesthetist in research team using protocol based
  1. insertion at mid-level of surgical insertion
  2. insertion depth is 3-5 cm in space, not more than 5 cm
  3. using benzoin tincture and transparent dressing to fix catheter
  4. test dose with 2%xylocaine with adrenaline 1:200,000 3ml If not cover desired dermatome: 2% lidocaine with adr added 3 ml every 5 min (up to 2 times)
  5. After induction and patients' hemodynamic are stable. Load 2 mg morphine with 0.0625% bupivacaine + morphine 0.02 mg/ml 3 ml then continuous infusion with rate according to initial local anesthetic requirement for incisional area coverage
  Arms: Protocol based

SUMMARY:
Epidural analgesia is the recommended analgesic technique in patients having surgery with severe postoperative pain such as thoracic and upper abdominal surgery. However, from the previous study, the incidence of inadequate pain control in patients receiving epidural analgesia is very high 48.6% in our hospital.

DETAILED DESCRIPTION:
A high incidence of inadequate epidural analgesia may result from variety of epidural techniques and epidural drug administrations. The protocol based practice has been developed from acute pain service which founded for more than 10 years. By using protocol based practice, the investigators believed that the incidence of inadequate epidural analgesia will be less compared with the current practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients age ≥ 18 years old undergo surgery with epidural catheter insertion at Siriraj hospital.

Exclusion Criteria:

* Coagulopathy
* Allergy to study drugs: local anesthetics and opioids
* History of chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Overall incidence of inadequate epidural analgesia | 72 hours
  To compare the overall incidence of inadequate epidural analgesia until considered removal between protocol-based and current practice by using the definition of inadequate analgesia as pain score of 4 or more out of 10 on numeric rating scale (0; no pain, 10; worst imaginable pain) at rest.

SECONDARY OUTCOMES:
Side effects | 72 hours
  To compare the incidence of undesirable side effects of epidural catheter between groups: sedation, respiratory depression, hypotension, motor weakness, postoperative nausea and vomiting and pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Pangthipampai, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No